CLINICAL TRIAL: NCT06688747
Title: Distal Versus Traditional Radial Access for Coronary Angiography and Intervention
Brief Title: The Primary Endpoint is to Compare the Incidence of Forearm RAO Between Distal and Traditional Radial Access Assessed by Vascular Ultrasound At Discharge
Acronym: RAO
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mostafa Talaat Bakr, Cardiology specialist, Assiut University
Other Study IDs: AssiutU/Mostafa Talaat
Record Dates: First submitted 2024-11-11; First posted 2024-11-14 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Coronary Angiography and Intervention
Keywords: RAO, DISTAL, Traditional radial
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Distal access: Distal radial access for coronary angiography and intervention
- Traditional access: Distal radial access for coronary angiography and intervention

SUMMARY:
The primary endpoint is to compare the incidence of forearm RAO between distal and traditional radial access for coronary angiography and intervention

DETAILED DESCRIPTION:
Trans radial access (TRA) has become the standard vascular access for coronary angiography and percutaneous coronary intervention (PCI) and is currently endorsed with a class IA recommendation in the latest European Society of Cardiology/European Association for Cardiothoracic Surgery (ESC/EACTS) Guidelines on myocardial revascularization, irrespective of clinical presentation Several clinical and procedural characteristics have been linked to the occurrence of RAO, and best practices recommendations for the prevention of RAO include reduction of the sheath/catheter size, adequate procedural anticoagulation, non-occlusive hemostasis (4) and a minimal pressure strategy with short (≤ 120 min) hemostasis time. The use of the distal radial artery with arterial access in the anatomical snuffbox or on the dorsum of the hand, has recently emerged as a promising alternative access route to further reduce the risk of RAO (5) The distal radial artery may be punctured proximally to the tendon of the extensor pollicis longus muscle in the anatomical snuffbox or distally to it in the dorsum of the hand.(6) the distal radial artery lies in the subcutaneous space superficial to the fascial compartments of the hand, thus favoring a faster, and safer hemostasis as compared to conventional TRA(7) The study will enroll 228 patients who will undergo a diagnostic coronary angiography and/or a PCI using a 6 Fr Sheath as the standard access sheath will be divided into two groups DRA versus TRA (114 cases in each group) The primary endpoint is the incidence of forearm RAO between the two groups at hospitalization discharge assessed by duplex ultrasound with independent investigator, who was not involved in the procedure. The presence or absence of a duplex ultrasound anterograde flow signal distal to the radial artery access site is checked between 8 to 48 hours post-procedure The secondary endpoints as successful sheath insertion, access site cross-over, total procedure time, sheath insertion time, puncture site bleeding overall bleeding, vascular access-site complication and radial artery spasm.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥18 y
2. Signed informed consent form
3. Indication to diagnostic coronary angiography or PCI
4. Patient's suitability for both DRA and conventional TRA using 6 Fr Sheath

Exclusion Criteria:

1. Chronic hemodialysis
2. Treatment of a coronary chronic total occlusion (CTO) lesion
3. Patients who underwent CA or PCI with radial access before

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will include patients will undergo coronary angiography and\or PCI in Assiut university heart hospital
Sampling Method: Probability Sample
Enrollment: 230 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
To compare the incidence of forearm RAO between distal and traditional radial access assessed by vascular ultrasound at discharge | One year
  The primary endpoint is the incidence of forearm RAO between the two groups at hospitalization discharge assessed by duplex ultrasound with independent investigator, who was not involved in the procedure. The presence or absence of a duplex ultrasound anterograde flow signal distal to the radial artery access site is checked between 8 to 48 hours post-procedure and follow up after 3 months

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sgueglia GA, Santoliquido A, Gaspardone A, Di Giorgio A. First Results of the Distal Radial Access Doppler Study. JACC Cardiovasc Imaging. 2021 Jun;14(6):1281-1283. doi: 10.1016/j.jcmg.2020.11.023. Epub 2021 Jan 13. No abstract available. PMID 33454250